CLINICAL TRIAL: NCT04982289
Title: A Phase 2a Randomized, Double-blind, Placebo-controlled, Parallel Groups, Multicenter Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of ALXN1830 Administered Subcutaneously in Adult Patients With Generalized Myasthenia Gravis
Brief Title: Study of ALXN1830 Administered Subcutaneously in Adults With Generalized Myasthenia Gravis
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor decision to terminate program
Sponsor: Alexion Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ALXN1830-MG-201
Record Dates: First submitted 2021-06-21; First posted 2021-07-29 (Actual); Last update posted 2022-02-11 (Actual); Status verified 2022-02

CONDITIONS: Generalized Myasthenia Gravis
Keywords: Generalized Myasthenia Gravis
MeSH Terms: conditions — Myasthenia Gravis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- ALXN1830 Dosing Arm 1 (Experimental): Participants will receive ALXN1830. Treatment will be received for 16 weeks followed by an Observation Period (no treatment) for 8 weeks.
  Interventions: Drug: ALXN1830
- ALXN1830 Dosing Arm 2 (Experimental): Participants will receive ALXN1830. Treatment will be received for 16 weeks followed by an Observation Period (no treatment) for 8 weeks.
  Interventions: Drug: ALXN1830
- ALXN1830 Dosing Arm 3 (Experimental): Participants will receive placebo for 8 weeks, then ALXN1830 for 8 weeks, followed by an Observation Period (no treatment) for 8 weeks.
  Interventions: Drug: ALXN1830; Other: Placebo

INTERVENTIONS:
Drug: ALXN1830 — Administered as an SC infusion.
Other: Placebo — Administered as an SC infusion.
  Arms: ALXN1830 Dosing Arm 3

SUMMARY:
This study will evaluate the safety, tolerability, pharmacokinetics and pharmacodynamics (PD), immunogenicity, and efficacy of subcutaneous (SC) ALXN1830 in adults with generalized myasthenia gravis (gMG).

DETAILED DESCRIPTION:
Participants have the option to enroll in an Open-label Extension (OLE) Period to receive ALXN1830 up to 58 weeks (including follow-up period).

ELIGIBILITY:
Key Inclusion Criteria:

* Diagnosis of myasthenia gravis.
* Positive serologic test for anti-acetylcholine receptor antibodies.
* Myasthenia Gravis Foundation of America Clinical Classification Class II to IV at Screening.
* MG-ADL profile must be ≥ 5.
* Participants receiving stable treatment with azathioprine; other immunosuppressive therapies.
* Total IgG level at Screening ≥ 600 milligrams/deciliter.

Key Exclusion Criteria:

* History of thymectomy, thymomectomy, or any other thymic surgery within 12 months prior to Screening.
* Any untreated thymic malignancy, carcinoma, or thymoma.
* Intravenous immunoglobulin within the 6 weeks, and/or use of plasmapheresis/plasma exchange prior to randomization (Day 1).
* Use of rituximab within the 3 months (90 days) prior to Screening.
* Participants who have received previous treatment with any biological agent or other anti-neonatal fragment crystallizable receptor therapy within 5 half-lives or 90 days after last dose (whichever is longer).
* Known medical or psychological condition(s) or risk factor that, in the opinion of the Investigator, might interfere with the participant's full participation in the study, pose any additional risk for the participant, or confound the assessment of the participant or outcome of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-01-01 (Estimated); Primary Completion 2023-01-31 (Estimated); Study Completion 2024-01-31 (Estimated)

PRIMARY OUTCOMES:
Adverse Events (AEs) And Serious Adverse Events (SAEs) Up To Week 24 | Up to Week 24
AEs And SAEs Up To Week 82 | Up to Week 82 (OLE)
Change From Baseline In Serum Total Immunoglobulin G (IgG) | Up to Week 24

SECONDARY OUTCOMES:
Change From Baseline In Myasthenia Gravis Activities Of Daily Living Profile (MG-ADL) Total Score | Up to Week 24
Change From Baseline In Quantitative Myasthenia Gravis (QMG) Score | Up to Week 24
Number Of Participants With At Least A 2-point Improvement In The MG-ADL Score Over 4 Consecutive Weeks | Up to Week 24
Number Of Participants With At Least A 3-point Improvement In The QMG Score Over 4 Consecutive Weeks | Up to Week 8
Change From Baseline In Neurological Disorders Fatigue Questionnaire (Neuro-Qol) Fatigue Score | Up to Week 24
Serum Trough Concentrations Of ALXN1830 | Up to Week 24
Change From Baseline In IgG Subtypes | Up to Week 24
Incidence Of Anti-drug Antibodies (ADA) And Neutralizing Antibodies (Nab) Against ALXN1830 | Up to Week 24
Titers Of ADA And Nab Against ALXN1830 | Up to Week 24

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Study Site, Phoenix, Arizona, United States